CLINICAL TRIAL: NCT05436899
Title: Training Simulator Efficacy in Developing Thoracic and General Surgical Skills in an Academic Residency Program: a Pilot Study
Brief Title: A Pilot Study on Training Simulator Efficacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Andrea Selenito Imperatori, Associate Professor of Thoracic Surgery, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LapSim training program
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Laparoscopic Surgery; Medical Education; Simulation Training
Keywords: Education; Simulation; Virtual reality; Laparoscopic surgery; Learning curve; Endoscopic surgery; Thoracoscopic surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive training group (Experimental): Participants in this group will undergo an intensive virtual training program twice a week
  Interventions: Other: LapSim training; Other: LapSim exam
- Non-Intensive training group (Active Comparator): Participants in this group will undergo a non-intensive virtual training program once a week
  Interventions: Other: LapSim training; Other: LapSim exam

INTERVENTIONS:
Other: LapSim training — Complete 4 courses, each of 12 weeks, of virtual reality simulation on LapSim surgical simulator.
Other: LapSim exam — Completed at the beginning and at the end of each of the 4 courses the corresponding exam task.

SUMMARY:
The purpose of this study is to plan an effective learning path in minimally invasive thoracic and general surgery with a virtual training simulator for trainees and to assess the improvement of residents' surgical skills by the introduction of this virtual training program.

DETAILED DESCRIPTION:
All thoracic and general surgery trainees at the first and second year of residency will be randomized in two groups: A) trainees undergoing an intensive (twice a week) virtual training program and B) those undergoing a non-intensive virtual training program (once a week).

The virtual training program will be organized in 4 modules, each of 12 weeks and, according to the training simulator instructions, for each surgical skill there are predetermined goals to be achieved by the trainee. Data about duration of surgical maneuvers and type and number of mistakes made by the trainee at each training session will be collected and compared with those of the same trainee at the previous session; this will assess the number of training sessions required to achieve the training simulator predetermined goals. Moreover, the same data will be registered at the beginning and at the end of each courses to compare the two groups of trainees (intensive vs non-intensive program).

ELIGIBILITY:
Inclusion Criteria:

* Trainees at the first and second year of residency in thoracic or general surgery

Exclusion Criteria:

* Fully trained surgeons
* Persons who are not trainees at year of specialization higher than the second

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Learning curves of time, errors and economy of motion for each training tasks | 48 weeks
  For each task, the computer automatically measures set parameters. Time, errors and economy of motion will be used in data analysis to create the learning curves for both intensive and non-intensive training group.

SECONDARY OUTCOMES:
Intensive vs non-intensive training group | 48 weeks
  For each exam tasks of the four training courses, compare the difference between the intensive and non-intensive training group, before and after each program training. Time, errors and economy of motion will be used in data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Imperatori, Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- Università degli Studi dell'Insubria, Varese, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data that underlie the results reported in this article (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Proposals should be directed to andrea.imperatori@uninsubria.it